CLINICAL TRIAL: NCT05737875
Title: DISPAIR vs. D-FRS - Establishing the Superiority of the Novel Distal Pancreatectomy Pancreatic Fistula Risk Prediction Models - A Multicenter International Retrospective Validation Study
Brief Title: Distal Pancreatectomy Pancreatic Fistula Risk Prediction Model Validation Study
Acronym: DPFValid
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: Helsinki University Central Hospital (Other); NHS Lothian, Royal Infirmary of Edinburgh (Unknown)
Responsible Party: Sponsor
Other Study IDs: DPFValid
Record Dates: First submitted 2023-02-10; First posted 2023-02-21 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Pancreatic Fistula; Pancreatectomy
MeSH Terms: conditions — Pancreatic Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Distal pancreatectomy: Patients who have undergone a distal pancreatectomy, retrospective analysis of post pancreatectomy fistula risk factors

SUMMARY:
Distal pancreas resection is a relatively rare procedure with a known risk of postoperative pancreatic fistula. Until quite recently, no valid risk prediction models for this have been available. In 2022 two different risk scores DISPAIR and D-FRS were published. The aim of this study is to compare, validate and possibly improve those scores in a international retrospective multicenter cohort.

DETAILED DESCRIPTION:
Fistula Risk Score (FRS) and its derivatives have been utilized in research surrounding pancreatoduodenectomy (Callery 2013, Mungroop 2019 & 2021). Distal pancreatectomy is a rare procedure, with typically less than 20 procedures a year performed by a large hepatopancreatobiliary surgery centre. A prediction model for pancreatic fistula after distal pancreatectomy had long been warranted and Ecker et al. were the closest at acquiring this in their 2019 study with over two thousand patients (Ecker 2019). However, not enough strongly associated variables were identified in their study to develop a prediction model. Very recently, two distinct models - the DISPAIR (Bonsdorff 2022) and the D-FRS (De Pastena 2022) - which both included pancreas-specific anthropometric measurements, were developed and validated. No studies comparing the performance of these models have been conducted and thus superiority of one model over other hasn't been established.

The DISPAIR relies on three preoperative variables: pancreatic thickness at the intended transection plane measured from preoperative CT-scans, site of transection (neck vs. body/tail) and history of diabetes. It was developed in 266 patients undergoing DP in Finland and externally validated with 402 patients from Sweden. It showed good discrimination and adequate calibration upon external validation with area under the curve (AUC) of 0.80, calibration intercept of 0.19 and slope of 0.72. The D-FRS is based on PT and main pancreatic duct (MPD) diameter at the pancreatic neck, both measured from preoperative CT-scans as well. It showed a satisfactory AUC of 0.73 after an internal-external validation procedure (Steyerberg 2016) where the development cohort of 339 patients was pooled with three distinct cohorts with a total sample size of 997 patients. Pooling validation cohort with the development cohort increases the optimism of model performance parameters, and strictly speaking does not count as a full external validation. The authors claimed D-FRS to be perfectly calibrated with a calibration intercept of 0 and slope of 1. Since this is in essence impossible, the soundness of the methodology behind the study is questionable (Van Calster 2019). Nonetheless, both models have identified similar novel risk factors for pancreatic fistula and show good potential for wider utilization.

The aim of this study is to compare and externally validate the performance of the DISPAIR and the D-FRS in a fully independent cohort of DP patients. The ultimate goal is to establish the potential superiority of one model over the other and identify directions for potential model updating.

As the DISPAIR is already externally validated we expect its performance to vary little and the AUC to set in the range of 0.75 - 0.85 in external validation cohorts. We expect to identify potential avenues of DISPAIR model updating with this external validation study. As the D-FRS has been validated with a pooled internal-external procedure it is more difficult to predict its performance but an AUC of over 0.70 would be expected.

The plan is to collect 200 patients per center, as this will give approximately 40 patients with a clinically relevant pancreatic fistula, allowing external validation and comparison of the scores center-wise also (in addition to pooled external validation and comparison).

ELIGIBILITY:
Inclusion Criteria:

* 18 to 99 years old
* Underwent distal pancreatectomy after 1/1/2020

Exclusion Criteria:

* Under 18 years old
* 100 years old or older
* Previous pancreatic surgery prior to distal pancreatectomy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have undergone a distal pancreatectomy
Sampling Method: Non-Probability Sample
Enrollment: 2284 (Actual)
Dates: Start 2023-04-07 (Actual); Primary Completion 2025-04-06 (Actual); Study Completion 2025-04-06 (Actual)

PRIMARY OUTCOMES:
Postoperative pancreatic fistula | 30 days postoperatively
  Postoperative pancreatic fistula

CONTACTS AND LOCATIONS:
Overall Officials: Ville Sallinen, MD PhD, Study Chair — Helsinki University Hospital and University of Helsinki; Stephen J Wigmore, MD FRCSED, Principal Investigator — University of Edinburgh
Locations (1):
- NHS Lothian, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plans for data sharing

REFERENCES:
- [Background] Callery MP, Pratt WB, Kent TS, Chaikof EL, Vollmer CM Jr. A prospectively validated clinical risk score accurately predicts pancreatic fistula after pancreatoduodenectomy. J Am Coll Surg. 2013 Jan;216(1):1-14. doi: 10.1016/j.jamcollsurg.2012.09.002. Epub 2012 Nov 2. PMID 23122535
- [Background] Mungroop TH, van Rijssen LB, van Klaveren D, Smits FJ, van Woerden V, Linnemann RJ, de Pastena M, Klompmaker S, Marchegiani G, Ecker BL, van Dieren S, Bonsing B, Busch OR, van Dam RM, Erdmann J, van Eijck CH, Gerhards MF, van Goor H, van der Harst E, de Hingh IH, de Jong KP, Kazemier G, Luyer M, Shamali A, Barbaro S, Armstrong T, Takhar A, Hamady Z, Klaase J, Lips DJ, Molenaar IQ, Nieuwenhuijs VB, Rupert C, van Santvoort HC, Scheepers JJ, van der Schelling GP, Bassi C, Vollmer CM, Steyerberg EW, Abu Hilal M, Groot Koerkamp B, Besselink MG; Dutch Pancreatic Cancer Group. Alternative Fistula Risk Score for Pancreatoduodenectomy (a-FRS): Design and International External Validation. Ann Surg. 2019 May;269(5):937-943. doi: 10.1097/SLA.0000000000002620. PMID 29240007
- [Background] Mungroop TH, Klompmaker S, Wellner UF, Steyerberg EW, Coratti A, D'Hondt M, de Pastena M, Dokmak S, Khatkov I, Saint-Marc O, Wittel U, Abu Hilal M, Fuks D, Poves I, Keck T, Boggi U, Besselink MG; European Consortium on Minimally Invasive Pancreatic Surgery (E-MIPS). Updated Alternative Fistula Risk Score (ua-FRS) to Include Minimally Invasive Pancreatoduodenectomy: Pan-European Validation. Ann Surg. 2021 Feb 1;273(2):334-340. doi: 10.1097/SLA.0000000000003234. PMID 30829699
- [Background] Ecker BL, McMillan MT, Allegrini V, Bassi C, Beane JD, Beckman RM, Behrman SW, Dickson EJ, Callery MP, Christein JD, Drebin JA, Hollis RH, House MG, Jamieson NB, Javed AA, Kent TS, Kluger MD, Kowalsky SJ, Maggino L, Malleo G, Valero V 3rd, Velu LKP, Watkins AA, Wolfgang CL, Zureikat AH, Vollmer CM Jr. Risk Factors and Mitigation Strategies for Pancreatic Fistula After Distal Pancreatectomy: Analysis of 2026 Resections From the International, Multi-institutional Distal Pancreatectomy Study Group. Ann Surg. 2019 Jan;269(1):143-149. doi: 10.1097/SLA.0000000000002491. PMID 28857813
- [Background] De Pastena M, van Bodegraven EA, Mungroop TH, Vissers FL, Jones LR, Marchegiani G, Balduzzi A, Klompmaker S, Paiella S, Tavakoli Rad S, Groot Koerkamp B, van Eijck C, Busch OR, de Hingh I, Luyer M, Barnhill C, Seykora T, Maxwell T T, de Rooij T, Tuveri M, Malleo G, Esposito A, Landoni L, Casetti L, Alseidi A, Salvia R, Steyerberg EW, Abu Hilal M, Vollmer CM, Besselink MG, Bassi C. Distal Pancreatectomy Fistula Risk Score (D-FRS): Development and International Validation. Ann Surg. 2023 May 1;277(5):e1099-e1105. doi: 10.1097/SLA.0000000000005497. Epub 2022 Jul 7. PMID 35797608
- [Background] Steyerberg EW, Harrell FE Jr. Prediction models need appropriate internal, internal-external, and external validation. J Clin Epidemiol. 2016 Jan;69:245-7. doi: 10.1016/j.jclinepi.2015.04.005. Epub 2015 Apr 18. No abstract available. PMID 25981519
- See also: Van Calster B, McLernon DJ, Van Smeden M, Wynants L, Steyerberg EW, Bossuyt P, et al. Calibration: The Achilles heel of predictive analytics. BMC Med. 2019;17(1):1-7. — https://doi.org/10.1186/s12916-019-1466-7